CLINICAL TRIAL: NCT03223428
Title: An Observational Study to Evaluate the Real-world Experience of Patients Who Are Initiating Treatment With Telotristat Ethyl (XERMELO™)
Brief Title: Real-world Evidence Study EvaLuating PAtient-Reported Outcomes With XERMELO
Acronym: RELAX
Status: Completed | Type: Observational
Sponsor: TerSera Therapeutics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: LX1606.1-401-CS; LX1606.401 (Other: TerSera Therapeutics)
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Carcinoid Syndrome
Keywords: neuroendocrine tumors, carcinoid syndrome, telotristat ethyl
MeSH Terms: conditions — Serotonin Syndrome; Neuroendocrine Tumors | interventions — telotristat ethyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carcinoid Syndrome patients initiating Xermelo: Patients with Carcinoid Syndrome who are initiating treatment with XERMELO.
  Interventions: Drug: Xermelo

INTERVENTIONS:
Drug: Xermelo — This study will include patients with carcinoid syndrome who are initiating treatment with XERMELO.
  Other Names: Telotristat ethyl

SUMMARY:
The primary objective of the study is to estimate the proportion of carcinoid syndrome (CS) patients who are satisfied with their overall symptom control, 6 months after initiating treatment with telotristat ethyl (XERMELO).

DETAILED DESCRIPTION:
This study will evaluate patient-reported outcomes for adults initiating telotristat ethyl (XERMELO) for carcinoid syndrome diarrhea (CSD) not adequately controlled by somatostatin analogs in US clinical practice. The primary objective is satisfaction with overall CS symptom control 6 months after starting XERMELO. Secondary objectives will evaluate satisfaction with control of CSD and flushing, CS symptoms, work productivity and activity impairment, SSA use, and weight. This study will provide real-world patient-reported outcomes in CS with XERMELO treatment for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult, ≥18 years of age at the time of informed consent
* A new, valid prescription for XERMELO
* Initiating XERMELO for the treatment of carcinoid syndrome
* Able and willing to provide informed consent prior to participation in the study

Exclusion Criteria:

* Unable to understand and read English
* Unable to access the internet
* Prior exposure to XERMELO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with CS and who are initiating treatment with XERMELO.
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janine North, BS, Study Director — TerSera Therapeutics LLC
Locations (1):
- RTI-HS, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li D, Darden C, Osman N, Sayeed S, Jackson L, Garbinsky D, Chauhan A. Real-World Clinical and Patient-Reported Outcomes from the Longitudinal Telotristat Ethyl Treatment Registry of Patients with Neuroendocrine Tumors. Cancer Manag Res. 2022 Oct 17;14:3009-3020. doi: 10.2147/CMAR.S386419. eCollection 2022. PMID 36262750
- See also: Prospective, observational, single-arm study evaluated long-term patient-reported outcomes in adults initiating TE in US clinical practice. The primary objective was satisfaction with overall CS symptom control at 6 months. — https://pubmed.ncbi.nlm.nih.gov/36262750/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were invited to participate in the RELAX study by the enrolling Specialty Pharmacies EnvoyHealth (also known as Diplomat Specialty Pharmacy and Optum Specialty Pharmacy) and Biologics Specialty Pharmacy.
Period: Overall Study
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Started | 223 (223 patients provided informed consent and completed baseline survey.)
Completed | 125 (125 Completed through Month 6 (primary endpoint))
Not Completed | 98
Not completed — No longer taking Xermelo | 27
Not completed — Declined Consent | 1
Not completed — Non-responders | 56
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Population: The analysis population will include all patients who provide consent, are enrolled into the study, and have data available for 1 or more of the primary and secondary endpoints.
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 223
Age, Categorical [Count of Participants; unit: Participants] — Population: Age was not collected for one (1) patient.
  Participants
    number analyzed (Participants) | 222
    <=18 years | 0
    Between 18 and 65 years | 138
    >=65 years | 84
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One patient did not provide age during the baseline survey
  years
    number analyzed (Participants) | 222
    (all) | 60.8 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 208
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 16
  White | 199
  More than one race | 4
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 223
Baseline Weight [Mean (Standard Deviation); unit: kilogram] — Weight collected in kilograms.
  kilogram | 80.9 (22.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are Satisfied With Their Overall Symptom Control
Description: The percentage of CS patients who are satisfied with their overall symptom control, 6 months after initiating treatment with telotristat ethyl (XERMELO). Satisfaction with how Xermelo has controlled diarrhea, flushing, and overall CS symptoms was assessed at the initial 6-month follow-up. The questionnaire allowed participants to choose a response on a 5-level Likert scale ranging from "Very dissatisfied" (level 1) to "Very satisfied" (level 5). For the assessments of satisfaction with control of diarrhea and flushing, "Not applicable" (level 0) was a response option for participants who do not have the particular symptom that is being assessed.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 125
Participants
  Very Satisfied with symptom control | 37
  Somewhat satisfied with symptom control | 58
  Neither satisfied or dissatisfied with symptom control | 22
  Somewhat dissatisfied with symptom control | 5
  Very dissatisfied with symptom control | 3

2. Secondary Outcome: Percentage of Patients Reporting Satisfaction of CS-related Diarrhea Control
Description: Estimate percentage of patients reporting satisfaction with CS-related diarrhea control from Baseline to 6 months after starting Xermelo. At baseline participants were asked, "Currently, how satisfied are you with how your diarrhea is controlled?" At the 6-month follow-up survey, participants were asked, "Currently, how satisfied are you with how Xermelo has controlled your diarrhea?"
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 125
Participants
  Very satisfied | 46
  Somewhat satisfied | 51
  Neither satisfied nor dissatisfied | 12
  Somewhat dissatisfied | 11
  Very dissatisfied | 5

3. Secondary Outcome: Percentage of Patients Reporting Satisfaction of CS- Related Flushing Control
Description: Estimate percentage of patients reporting satisfaction with CS-related flushing control from Baseline to 6 Months. At baseline, participants who had reported flushing as a symptom were asked, "Currently, how satisfied are you with how your flushing is controlled?" At 6 months, participants who had reported flushing as a symptom at Baseline were asked, "Currently, how satisfied are you with how Xermelo has controlled your flushing?"
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 108
Participants
  Very satisfied | 24
  Somewhat satisfied | 39
  Neither satisfied nor dissatisfied | 34
  Somewhat dissatisfied | 7
  Very dissatisfied | 4

4. Secondary Outcome: Number of Patients Reporting Reduction in Rescue SSA Use
Description: Number of participants reporting a reduction in rescue SSA use at 6 months after initiating treatment with Xermelo.
Time Frame: Baseline to 6 months
Measure: Number; unit: participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 104
participants | 21

5. Secondary Outcome: Percentage of Patients Reporting Reduction in the Dose of Long-acting SSA Injection
Description: Percentage of patients reporting a reduction in the dose of long-acting SSA injection 6 months after patients initiated treatment with Xermelo
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 125
Participants | 7

6. Secondary Outcome: Percentage of Patients Reporting Reduction in the Frequency of Long-acting SSA Injection
Description: Estimate Percentage of Patients Reporting Reduction in the Frequency of Long-acting SSA Injection 6 months after patients initiated treatment with Xermelo
Time Frame: Baseline to 6 months
Population: There was a discrepancy between how many patients answered the survey for "Reduction in dose of long-acting SSA" (n=125) and "Reduction in frequency of long-acting SSA" (n=123). Two people did not answer the latter question but did answer the former.
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 123
Participants | 9

7. Secondary Outcome: Percentage of Patients Reporting an Overall Improvement in CS Symptom Control Based on Patient Global Impression of Change (PGIC)
Description: Estimate percentage of patients reporting an overall improvement in CS symptom control (diarrhea, flushing, frequency of BMs) after initiating Xermelo based on Patient Global Impression of Change (PGIC)
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 125
Participants
  Very much improved | 20
  Much improved | 28
  Somewhat improved | 49
  No change | 20
  Somewhat worse | 6
  Much worse | 1
  very much worse | 1

8. Secondary Outcome: Percentage Change of Patients Who Had Reduction in Work-related Absenteeism, Presenteeism, Activity Impairment, and Overall Productivity Loss From Baseline to 6 Months After Initiating Telotristat Ethyl Based on WPAI-SHP
Description: Estimate of the percentage of patients who had reduction in work-related absenteeism, presenteeism, activity impairment, and overall productivity loss based on Worker Productivity and Activity Impairment: Specific Health Problem v2.0 (WPAI- SHP). The percentage change was measured from baseline to 6 months after treatment with telotristat ethyl.
Time Frame: Baseline to 6 months
Population: Only 124 patients answered the work activity and impairment questionnaire. Not all patients were employed and only a small subset were eligible to answer the Absenteeism, Presenteeism and Work Productivity Loss. Only 34, 32 and 32 patients answered those questionnaires, respectively.
Measure: Mean (Standard Deviation); unit: percentage change baseline to Month 6
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 125
percentage change baseline to Month 6
  Absenteeism: number analyzed (Participants) | 34
  Absenteeism | 4.1 (21.86)
  Presenteeism: number analyzed (Participants) | 32
  Presenteeism | -9.7 (20.76)
  Work productivity loss: number analyzed (Participants) | 32
  Work productivity loss | -10.1 (19.60)
  Activity impairment: number analyzed (Participants) | 124
  Activity impairment | -8.1 (26.86)

9. Secondary Outcome: Percentage of Patients Reporting Weight Gain
Description: Estimate of the percentage of patients reporting weight gain after initiating Xermelo therapy.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
Number analyzed (Participants) | 125
Participants | 24

ADVERSE EVENTS:
Time Frame: Adverse events not collected as part of the survey.
Description: All-cause mortality, serious and other (not serious) adverse events were not collected or assessed during this study.
Arm/Group | Carcinoid Syndrome Patients Initiating Xermelo
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
A potential for responder bias was possible as results were self-reported. Decreased number of responders presented challenges to interpretation after approx. 24-30 months, hence findings should be interpreted with caution.

Adverse event safety data collection: Out of scope of this study. Reported adverse events, if occurred, were to be collected and reported to the Sponsor outside of the survey collection process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT03223428/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03223428/SAP_001.pdf